CLINICAL TRIAL: NCT06432647
Title: ATH-1105 A Phase 1, Double-Blind, Placebo-Controlled, Single-and-Multiple-Oral-Dose, Safety, Tolerability, and Pharmacokinetic Study in Healthy Male and Female Subjects
Brief Title: A SAD and MAD Study of the Safety, Tolerability, and Pharmacokinetics of ATH-1105
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athira Pharma (Industry)
Collaborators: Fortrea Holdings, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: ATH-1105-0101
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
Keywords: ATH-1105

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ATH-1105 (Experimental): Part A: ATH-1105 administered once as an oral solution.
  Part B: ATH-1105 administered once daily as an oral solution for 10 days.
  Interventions: Drug: ATH-1105
- Placebo (Placebo Comparator): Part A: Placebo administered once as an oral solution
  Part B: Placebo administered once daily as an oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH-1105 — ATH-1105 in oral form. Participants will be administered ATH-1105 once in Part A and once daily for 10 days in Part B.
  Arms: ATH-1105
Drug: Placebo — Placebo in oral form. Participants will be administered Placebo once in Part A and once daily for 10 days in Part B.
  Arms: Placebo

SUMMARY:
The goal of this Phase 1 interventional study is to assess the safety, tolerability and pharmacokinetics of ATH-1105 in healthy male and female participants.

DETAILED DESCRIPTION:
The study is a Phase 1, First-In-Human study consisting of two parts (A and B). Part A will comprise a single-dose, double-blind, placebo-controlled, sequential-group design. Part B will comprise a multiple-dose, placebo-controlled, sequential-group design.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2 inclusive.
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations at screening and check-in or predose on Day 1
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

Medical Conditions:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* Any of the following:

  1. QTcF >450 ms in males or >470 ms in females
  2. QRS duration >110 ms
  3. PR interval >220 ms
  4. Findings which would make QTc measurements difficult or QTc data uninterpretable.
  5. History of additional risk factors for torsades de pointes
* Confirmed systolic blood pressure >140 or <90 mmHg, diastolic blood pressure >90 or <50 mmHg, and pulse rate >100 or <40 beats per minute.
* Positive hepatitis panel and/or positive human immunodeficiency virus test
* Part B only: Current psychiatric disorder, suicidal ideation in the previous 2 years (as assessed by the Columbia-Suicide Severity Rating Scale [C-SSRS]), or a lifetime suicide attempt.

Prior/concomitant therapy:

* Administration of any vaccine in the 30 days prior to dosing.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes
* Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing
* Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to check-in

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Part A: Up to 7 days post-dose, Part B: Up to 7 days post final dose on day 10
  Safety and tolerability of single or multiple ascending doses of ATH-1105 as measured by incidence of AEs, determined by clinical laboratory tests, physical examinations, vital signs measurements, and 12-lead ECG
Severity of Treatment-Emergent Adverse Events | Part A: Up to 7 days post-dose, Part B: Up to 7 days post final dose on day 10
  Treatment-emergent adverse events will be graded on a 1 through 5 scale, based on severity as determined by the principal investigator.

SECONDARY OUTCOMES:
Area under the plasma concentration time curve (AUC) | Part A: Up to 48 hours post-dose, Part B: Up to 48 hours post final dose on Day 10
  AUC will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Maximum observed plasma concentration (Cmax) | Part A: Up to 48 hours post-dose, Part B: Up to 48 hours post final dose on Day 10
  Cmax will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Time to maximum observed plasma concentration (Tmax) | Part A: Up to 48 hours post-dose, Part B: Up to 48 hours post final dose on Day 10
  Tmax will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Half-life (t1/2) | Part A: Up to 48 hours post-dose, Part B: Up to 48 hours post final dose on Day 10
  t1/2 will be determined from all collected plasma samples from baseline through up to 48 hours post-dose.
Amount of IMP excreted unchanged in the urine (Ae) | Part A: Up to 48 hours post-dose, Part B: Up to 48 hours post final dose on Day 10
  Amount of IMP excreted unchanged in the urine will be determined from all collected urine samples from baseline through up to 48 hours post-dose
IMP Concentration in Cerebrospinal Fluid | Will occur at calculated maximum plasma concentration.
  Amount of IMP in the urine will be determined from all collected CSF samples from baseline through up to 48 hours post-dose
Accumulation Ratio (AUC) of IMP in Urine | Part A: Up to 48 hours post-dose, Part B: Up to 48 hours post final dose on Day 10
  Accumulation Ratio in urine will be determined from all collected urine samples from baseline through up to 48 hours post-dose
Accumulation Ratio (AUC) of IMP in Plasma | Part A: Up to 48 hours post-dose, Part B: Up to 48 hours post final dose on Day 10
  Accumulation Ratio in plasma will be determined from all collected plasma samples from baseline through up to 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea Clinical Research Unit Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No